CLINICAL TRIAL: NCT01973101
Title: Phase II, Prospective, Randomized, Non-comparative Study of Treatment With Induction Chemotherapy With Cisplatin and Gemcitabine Followed by Chemoradiation or Definitive Chemoradiation in Invasive Locally Advanced Carcinomas of Uterine Cervix.
Brief Title: Non-comparative Study of Treatment With Induction Chemotherapy With Cisplatin and Gemcitabine Followed by Chemoradiation or Definitive Chemoradiation in Invasive Locally Advanced Carcinomas of Uterine Cervix.
Acronym: CIRCE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP 217/2012
Record Dates: First submitted 2013-10-22; First posted 2013-10-31 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Patients Diagnosed With Advanced Carcinoma of Uterine Cervix t
Keywords: Advanced carcinomas of uterine cervix; Chemoradiation; Chemo-induction; Cisplatin; Gemcitabine
MeSH Terms: interventions — Cisplatin; Gemcitabine; Radiotherapy; Brachytherapy

ARMS (2):
- Chemo-induction (Experimental): Cisplatin plus Gemcitabine for 3 cycles followed by Cisplatin, radiotherapy and brachytherapy
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Radiation: Radiotherapy; Radiation: Brachytherapy
- Chemoradiotherapy (Active Comparator): Cisplatin, radiotherapy and brachytherapy
  Interventions: Drug: cisplatin; Radiation: Radiotherapy; Radiation: Brachytherapy

INTERVENTIONS:
Drug: Cisplatin — 50 mg/m2 - Day 1
  Arms: Chemo-induction
Drug: Gemcitabine — Gemcitabine 1000mg/m2 on day 1 and day 8.
  Arms: Chemo-induction
Drug: cisplatin — Cisplatin 40 mg/m2 on day 1, day8, day15, day22, day 36 of radiotherapy period.
Radiation: Radiotherapy — 45 Gy
Radiation: Brachytherapy — 80 Gy

SUMMARY:
The purpose of this phase II study is to determine the survival free disease of patients diagnosed with invasive locally advanced carcinomas of uterine cervix treated with induction chemotherapy with cisplatin and gemcitabine followed by chemoradiation and definitive chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced carcinoma of uterine cervix histological confirmed.
2. Indication for definitive chemoradiation treatment;
3. Measurable disease by RECIST 1.1 (Response Evaluation Criteria in Solid Tumors) criteria;
4. Age between 18 years old and 70 years old;
5. Adequate bone marrow and organ function defined by laboratory values;
6. Non evidence of disease in para-aortic lymph node;

Exclusion Criteria:

1. Previous treatment with Chemotherapy or radiotherapy
2. Previous surgery for primary tumor;
3. Distant metastasis;
4. Performance status according to Eastern Cooperative Oncology Group greater than 2;
5. Peripheric neuropathy greater than grade 2 by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE) version 3.0;
6. Significant Cardiac disease (history of and/or active disease);
7. Other treatment for cancer, including hormonotherapy;
8. Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements;

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-06; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | From the randomization until the end of the treatment - up to 36 month.

SECONDARY OUTCOMES:
Response rate | 36 month after the end of the treatment.
Locoregional disease control rate | 36 month after the end of treatment.
Acute and chronic toxicity in both arms | From the randomization until the end of the treatment.
Overall survival | 36 month after the end of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Del Pilar Estevez Diz, MD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- ICESP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Nunes de Arruda F, da Costa S, Bonadio R, Dornellas A, Pereira D, de Bock GH, Del Pilar Estevez Diz M. Quality of life of locally advanced cervical cancer patients after neoadjuvant chemotherapy followed by chemoradiation versus chemoradiation alone (CIRCE trial): a randomized phase II trial. Int J Gynecol Cancer. 2020 Jun;30(6):749-756. doi: 10.1136/ijgc-2019-001134. Epub 2020 Apr 21. PMID 32321767
- [Derived] da Costa SCS, Bonadio RC, Gabrielli FCG, Aranha AS, Dias Genta MLN, Miranda VC, de Freitas D, Abdo Filho E, Ferreira PAO, Machado KK, Scaranti M, Carvalho HA, Estevez-Diz MDP. Neoadjuvant Chemotherapy With Cisplatin and Gemcitabine Followed by Chemoradiation Versus Chemoradiation for Locally Advanced Cervical Cancer: A Randomized Phase II Trial. J Clin Oncol. 2019 Nov 20;37(33):3124-3131. doi: 10.1200/JCO.19.00674. Epub 2019 Aug 26. PMID 31449470